CLINICAL TRIAL: NCT06894823
Title: Development of a Platform for the Clinical Implementation of Precision Oncology in the Central-Southern Regions of Italy (COESIT)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: COESIT
Record Dates: First submitted 2025-03-13; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Creation of a laboratory network — Creation of a laboratory network in Central-Southern Italy capable of performing complex genomic analyses.
Other: Mapping of genomic alterations — Mapping of genomic alterations aimed at precision medicine and personalized diagnostic and therapeutic approaches.
Other: Creation of a bioinformatics network among the participating institutions. — Creation of a bioinformatics network among the participating institutions.
Other: Development of a platform for the collection of clinicopathological and genetic-molecular data. — Development of a platform for the collection of clinicopathological and genetic-molecular data.
Other: Identification of prognostic and predictive factors for the implementation of precision oncology strategies based on genomic profiling. — Identification of prognostic and predictive factors for the implementation of precision oncology strategies based on genomic profiling.

SUMMARY:
COESIT aims to establish a network of reference laboratories in the central-southern regions of Italy for the genetic and molecular characterization of tumors, with the goal of implementing precision and personalized oncology in clinical practice.

DETAILED DESCRIPTION:
The project will begin with a technological upgrade of the laboratories and the standardization of sequencing procedures and bioinformatics analyses, involving all institutions participating in the initiative. Subsequently, a shared database will be created, integrating sequencing data and clinicopathological information. This will enable research projects aimed at expanding knowledge on the genetic alterations of tumors in patients from central-southern Italy and identifying prognostic and predictive biomarkers that support the implementation of precision and personalized medicine.

The enhancement of genomic laboratories, the sharing of analytical procedures and bioinformatics protocols, and the development of a common database of sequencing and clinicopathological data will serve as essential tools to deepen specific knowledge on the genomic characteristics of tumors in patients from southern Italy. This will facilitate the clinical implementation of precision and personalized medicine based on genomic analysis.

The study is multicentric and observational. The nature of the data included will be both retrospective and prospective, as described below:

1. Prospective collection of clinicopathological information, including lifestyle factors and exposure to environmental and occupational carcinogens, as well as CGP (Comprehensive Genomic Profiling) data obtained through targeted sequencing techniques. These data will be generated within clinical practice or local genomic screening programs, with the patient's informed consent.
2. Analysis of the correlation between tumor heterogeneity-specifically genomic biomarkers-and therapy response in all enrolled patients who did not respond to targeted therapy administered according to current clinical guidelines.
3. Retrospective collection of clinicopathological information and CGP data from case series available in COESIT center biobanks for the identification of new biomarkers. Specific sub-studies will be proposed with amendments to the main study described here.
4. Collection of information on germline alterations in individuals at risk for breast and gastric cancer, already analyzed within approved protocols , with the subject's informed consent for data inclusion in the COESIT platform.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Patients from the central-southern regions

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients from the central-southern regions of Italy diagnosed with lung, breast, colorectal, ovarian, liver, bile duct, pancreatic, and gastric cancers.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of diagnostic precision in oncology based on advanced molecular profiling tools. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonella De Luca, Principal Investigator — Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale
Locations (1):
- Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale, Napoli, Italy